CLINICAL TRIAL: NCT03905421
Title: Quality of Life Assessed With the PAH SYMPACT Questionnaire in the Pulmonary Hypertension Clinic
Brief Title: Quality of Life Assessed With the PAH SYMPACT Questionnaire
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hilary M. DuBrock, MD, Principal Investigator, Mayo Clinic
Other Study IDs: 19-000630
Record Dates: First submitted 2019-03-13; First posted 2019-04-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- usual care: The patient will be seen in the PH clinic and will be approached to consent and participate in the SYMPACT trial. They will not be randomized to palliative care.
- palliative care: The patient will be seen in the PH clinic and will be approached to consent and participate in the SYMPACT trial. Based on the patients in Group 1 and 3 PH and a high SYMPACT score> 1.0 in any domain they will be randomized to receive standard care or a palliative care initial consult.

SUMMARY:
Researchers are evaluating quality of life in pulmonary hypertension subjects using the Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire and assessing the questionnaires' performance with regard to relationship to other markers of disease severity, response to treatment, and outcome in a clinical practice setting.

DETAILED DESCRIPTION:
Subjects will be recruited from among those seen at the Mayo Pulmonary Hypertension Clinic. The PAH-SYMPACT questionnaire will be administered either in written form or by telephone interview.

On the second 100 patients implement a standardized palliative care referral program for patients with Group 1 and 3 PH and high SYMPACT scores> 1.0.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Consents to participate
* Documented group I PAH based upon these hemodynamic criteria: (mPAP > 20, PCW 18 or less, PVR > 3 Wood units
* Mean PAP > 20, PCW ≤ 18, PVR > 3 Wood units
* Parenchymal lung disease that in the opinion of the investigator qualifies patient as group III PH
* Documented chronic thromboembolic pulmonary hypertension or chronic thromboembolic disease with intent to treat with surgery, balloon pulmonary angioplasty, and/or PH medication

Exclusion Criteria:

* Left sided heart disease (LVEF<50%, PAWP>18)
* Any other known concomitant life-threatening disease with a life expectancy <12 months
* Any other clinically relevant and/or serious chronic medical condition that would affect study participation in the opinion of the investigator
* Non English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from among those seen at the Mayo Pulmonary Hypertension Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Quality of life in pulmonary hypertension subjects | Baseline
  Measured using the Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire using a scale of 0=no, 1=mild, 2=moderate, 3=severe, and 4=very severe
Quality of life in pulmonary hypertension subjects | 14 months
  Measured using the Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire using a scale of 0=no, 1=mild, 2=moderate, 3=severe, and 4=very severe

CONTACTS AND LOCATIONS:
Overall Officials: Hilary M DuBrock, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No